CLINICAL TRIAL: NCT02361736
Title: Evaluate the Nephrotoxicity by 6% Hydroxyethyl Starch 130/0.4 in Old Patients
Brief Title: Evaluate the Nephrotoxicity by 6% Hydroxyethyl Starch 130/0.4 in Old Patients During Orthopaedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuanyuan Zhang (Other)
Collaborators: Tianjin Union Medical Center (Other); Tianjin First Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Yuanyuan Zhang, Tianjin Medical University General Hospital Ethics Committee, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: IRB2014-102-01
Record Dates: First submitted 2015-02-02; First posted 2015-02-12 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Total Fluid Volume Increased
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactate Ringers (Sham Comparator): Lactate Ringers is intravenously administrated at a dose of 7.5ml/kg during the surgery
  Interventions: Drug: Lactate Ringers
- Hydroxyethyl Starch (Experimental): 6% Hydroxyethyl Starch (HES) is intravenously administrated at a dose of 7.5ml/ kg in the first hour of surgery, and then, Lactate Ringers' is administrated to the patient until the end of the surgery
  Interventions: Drug: Hydroxyethyl Starch

INTERVENTIONS:
Drug: Hydroxyethyl Starch — 6% Hydroxyethyl Starch(HES) is intravenously given 7.5ml/kg for the first hour of surgery
  Other Names: HES
  Arms: Hydroxyethyl Starch
Drug: Lactate Ringers — Lactate Ringers is intravenously administrated at a dose of 7.5ml/kg during the surgery
  Other Names: LR
  Arms: Lactate Ringers

SUMMARY:
Hydroxyethyl starch (HES) is commonly used as plasma expander during surgery but may be nephrotoxic as seen in studies in patients with sepsis. The investigators hypothesized that the possible nephrotoxicity of 6% HES 130/0.4 could be revealed by measurements of urinary and plasma neutrophil gelatinase-associated lipocalin and interleukin-18 (IL-18) in old patients with normal renal function during orthopaedic surgery.

DETAILED DESCRIPTION:
Hydroxyethyl starch (HES) is widely used as volume expander to maintain circulation in patients during surgery, trauma, and in critical disease, where a rapid and sustained volume expansion is the goal. However, acute kidney injury (AKI) is sometimes a complication in these patients and HES might be a contributing factor. Acute kidney injury is often diagnosed using a sudden rise in plasma creatinine (p-crea) or an abrupt decrease in urine output. P-crea depends on sex, nutrition, medication,muscle mass, and age and it increases 24 to 48 h after renal injury, so the diagnosis of AKI is delayed when using p-crea alone as an indicator for renal damage. New technology allows for earlier diagnosis of AKI using measurements of biomarkers in urine. Neutrophil gelatinase-associated lipocalin (NGAL) is a small protein, which is filtered via the glomeruli and reabsorbed in the proximal tubules, and thus low concentrations of NGAL can be measured in the blood and urine. Approximately 6 h after a renal injury, NGAL increases rapidly due to an up-regulated expression and secretion in the epithelial cells of the thick ascending limb of Henle's loop, the distal tubules, and the collecting ducts. Thus, NGAL can be used as a marker of renal damage. However, infections and malignancies can give falsely increased levels.

Interleukin-18 (IL-18) is mainly created from proximal kidney tubules which is a proinflammatory factor that can be detected in earlier urine of AKI animal models. There is significant rise in IL-18 levels in urine of AKI confirmed cases(no chronic kidney disease, no urinary tract infections, no prerenal factors), specificity and susceptibility is 90%. As a result, IL-18 can be selected as a biomarker.

Intravenously administrated HES is excreted in urine but is also partly accumulated in the tissues. Studies in animals and humans showed that HES molecules were accumulated in the proximal tubule cells with subsequent vacuolization and swelling-a condition known as osmotic nephrosis. However, recent studies, primarily conducted in patients with sepsis, found impaired renal function even when using tetrastarch. In contrast, perioperative studies found no evidence of AKI after infusion of HES. The investigators hypothesized that 6% HES 130/0.4 had a nephrotoxic effect, which could be revealed by measurements of urinary and plasma NGAL and IL-18; that 6% HES 130/0.4 influenced kidney function differently than crystalloids(lactated Ringer's solution) due to the different pharmacokinetic properties of colloids compared with that of crystalloids.

ELIGIBILITY:
Inclusion Criteria:

* Old patients scheduled to undergo orthopaedic surgery under a intravertebral anesthesia. (American Society of Anesthesiologists physical status I-Ⅲ)

Exclusion Criteria:

* Allergy and contraindication to HES
* Infections and malignancies
* Sepsis
* History of heart failure or New York Heart Association(NYHA)>Ⅲ
* Renal failure or Cr>108μmol/L，BUN>8.3mmol/L
* Undergoing dialytic treatments
* Intracranial hemorrhages
* Taking non-steroidal antiinflammatory agent for a long time
* Inability to understand the Study Information Sheet and provide a written consent to take part in the study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Yonghao, M.D.,Ph.D, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Y, Yu Y, Jia J, Yu W, Xu R, Geng L, Wei Y. Administration of HES in elderly patients undergoing hip arthroplasty under spinal anesthesia is not associated with an increase in renal injury. BMC Anesthesiol. 2017 Feb 21;17(1):29. doi: 10.1186/s12871-017-0320-8. PMID 28222674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2015 to January 2016, patients were recruited and estimated for eligibility.
Pre-assignment Details: Exclusion criteria:Allergy and contraindication to HES; Infections and malignancies; Sepsis; History of heart failure or NYHA>Ⅲ; Renal failure or Cr>108μmol/L，BUN>8.3mmol/L;Undergoing dialytic treatments; Intracranial hemorrhages;Taking non-steroidal antiinflammatory agent for a long time
Period: Overall Study
Arm/Group | Lactate Ringers | Hydroxyethyl Starch
Started | 60 | 60
Completed | 59 | 59
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Ages Eligible for Study: ≥65 Years； Both Genders；No Healthy Volunteers
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactate Ringers | Hydroxyethyl Starch | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: age] | 76.4 (8.1) | 75.9 (7.5) | 76.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Concentration of NGAL in Urine on 5 Time Point
Description: Neutrophil gelatinase-associated lipocalin (NGAL) is a small protein, which is filtered via the glomeruli and reabsorbed in the proximal tubules, and thus low concentrations of NGAL can be measured in the blood and urine.
Time Frame: -1d, 0d, 1d, 3d, 5d after surgery
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lactate Ringers | Hydroxyethyl Starch
Number analyzed (Participants) | 59 | 59
ng/ml
  -1d | 5.6 (0.7) | 4.9 (0.8)
  0d | 5.2 (0.4) | 5.1 (0.3)
  1d | 4.9 (0.3) | 4.9 (0.4)
  3d | 5.0 (0.3) | 5.2 (0.5)
  5d | 4.3 (0.8) | 5.1 (0.4)

2. Primary Outcome: Concentration of IL-18 in Urine on 5 Time Point
Description: IL-18 is mainly created from proximal kidney tubules which is a proinflammatory factor that can be detected in earlier urine of AKI animal models.
Time Frame: -1d, 0d, 1d, 3d, 5d after surgery
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Lactate Ringers | Hydroxyethyl Starch
Number analyzed (Participants) | 59 | 59
μg/L
  -1d | 86.6 (8.5) | 82.7 (8.5)
  0d | 83.2 (4.8) | 89.5 (5.8)
  1d | 118.5 (11.4) | 109.6 (9.2)
  3d | 142.6 (18.1) | 140.5 (10.9)
  5d | 162.0 (18.5) | 159.7 (16.9)

3. Primary Outcome: Concentration of IL-18 in Plasma on 5 Time Point
Time Frame: -1d, 0d, 1d, 3d, 5d after surgery
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Lactate Ringers | Hydroxyethyl Starch
Number analyzed (Participants) | 59 | 59
μg/L
  -1d | 81.0 (14.5) | 79.3 (9.8)
  0d | 81.4 (9.0) | 81.0 (10.4)
  1d | 83.8 (12.5) | 84.2 (13.8)
  3d | 86.5 (14.1) | 83.4 (10.2)
  5d | 81.5 (6.1) | 85.1 (11.3)

4. Secondary Outcome: Concentration of β2 Microglobulin in Urine
Time Frame: -1d, 0d, 1d, 3d, 5d after surgery
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Lactate Ringers | Hydroxyethyl Starch
Number analyzed (Participants) | 59 | 59
mg/L
  -1d | 93.2 (8.9) | 96.4 (11.2)
  0d | 90.6 (8.2) | 97.1 (12.2)
  1d | 99.8 (14.2) | 101.7 (9.4)
  3d | 104.7 (15.0) | 99.4 (15.7)
  5d | 93.2 (12.3) | 103.0 (13.8)

5. Secondary Outcome: Estimated Glomerular Filtration Rate(eGFR) on 5 Time Point
Description: eGFR is calculated by concentration of creatinine and CKD-EPI2009
Time Frame: -1d, 0d, 1d, 3d, 5d after surgery
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Lactate Ringers | Hydroxyethyl Starch
Number analyzed (Participants) | 59 | 59
mL/min/1.73m2
  -1d | 61.9 (8.3) | 63.9 (14.3)
  0d | 63.5 (9.6) | 63.5 (13.5)
  1d | 63.0 (6.2) | 64.0 (14.4)
  3d | 64.0 (9.4) | 72.8 (10.4)
  5d | 66.4 (9.2) | 68.6 (12.4)

6. Primary Outcome: Concentration of NGAL in Plasma on 5 Time Point.
Description: concentration of NGAL in plasma on 5 time point. Biomarkers are measured by ELISA.
Time Frame: -1d, 0d, 1d, 3d, 5d after surgery
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lactate Ringers | Hydroxyethyl Starch
Number analyzed (Participants) | 59 | 59
ng/ml
  -1d | 4.1 (0.8) | 4.0 (0.3)
  0d | 4.0 (0.7) | 4.2 (0.5)
  1d | 4.4 (0.9) | 4.3 (0.5)
  3d | 4.1 (0.7) | 4.2 (0.5)
  5d | 4.3 (0.8) | 4.4 (0.6)

7. Secondary Outcome: Ratio of the Urine Trace Albumin and Creatinine(ACR) on 5 Time Point
Description: ACR is calculated by the urine trace albumin divided by the urine creatinine
Time Frame: -1d, 0d, 1d, 3d, 5d after surgery
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lactate Ringers | Hydroxyethyl Starch
Number analyzed (Participants) | 59 | 59
ratio
  -1d | 1.89 (0.14) | 1.96 (0.21)
  0d | 1.84 (0.20) | 1.98 (0.19)
  1d | 1.90 (0.19) | 1.90 (0.09)
  3d | 1.94 (0.15) | 1.99 (0.13)
  5d | 1.92 (0.12) | 1.95 (0.20)

ADVERSE EVENTS:
Arm/Group | Lactate Ringers | Hydroxyethyl Starch
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

LIMITATIONS AND CAVEATS:
We may have to prolong the follow-up visit for patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes